CLINICAL TRIAL: NCT02263157
Title: Evaluate the Association Between Blood Stream Infection (BSI) and Thrombocytopenia (Surgical Intensive Care Unit)SICU Patients
Brief Title: Evaluate the Association Between Infection and Thrombocytopenia
Status: Completed | Type: Observational
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Jianan Ren, BSI-PLT, Jinling Hospital, China
Other Study IDs: BSI-PLT
Record Dates: First submitted 2014-10-05; First posted 2014-10-13 (Estimated); Last update posted 2014-10-13 (Estimated); Status verified 2014-10

CONDITIONS: Thrombocytopenia
MeSH Terms: conditions — Thrombocytopenia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (4):
- BSI group with thrombocytopenia: BSI patients with thrombocytopenia
- Non-BSI group with thrombocytopenia: Non-BSI patients with thrombocytopenia
- BSI group without thrombocytopenia: BSI patients without thrombocytopenia
- Non-BSI group without thrombocytopenia: Non-BSI patients without thrombocytopenia

SUMMARY:
The study is designed to evaluate the association between nosocomial bloodstream infection and the occurrence of thrombocytopenia in surgical critical ill patients.

ELIGIBILITY:
Inclusion Criteria:

* Sequential consenting adult patients of either sex were prospectively enrolled into the study.

Exclusion Criteria:

* Patients who passed away within 24 hours after hospitalization would be excluded.

Patients who developed into a bloodstream infection within 48 hours after hospital admission were also excluded.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sequential consenting adult patients of either sex were prospectively enrolled into the study.
Sampling Method: Non-Probability Sample
Enrollment: 390 (Actual)
Dates: Start 2013-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
mortality rate | 28 days